CLINICAL TRIAL: NCT01538238
Title: pazopanib_NCRCC,Ph2 STUDY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ho Yeong Lim, Professor of Medicine, Sungkyunkwan University School of Medicine, Department of Hematology and Oncology, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-01-056
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Locally Advanced or Metastatic Non-clear Cell Type Renal Cell Carcinoma
MeSH Terms: interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pazopanib (Experimental): pazopanib 800mg qd
  Interventions: Drug: pazopanib

INTERVENTIONS:
Drug: pazopanib — pazopanib 800mg qd until progression or unacceptable toxicity

SUMMARY:
Recent advances in understanding the biology and genetics of renal cell carcinoma (RCC) have led to major therapeutic implications. Von Hippel-Lindau (VHL) gene inactivation, present in the majority of sporadic forms of RCC, leads to a defective VHL protein, followed by an active transcription of hypoxia-inducible genes, including vascular endothelial growth factor (VEGF), platelet-derived growth factor (PDGF), c-kit, and others. However, the concept of VHL inactivation in RCC and the subsequent malignant phenotype is almost exclusively seen in patients with clear cell histology.

The data about efficacy of VEGF receptor inhibitors for non-clear cell RCC (NCRCC) is rare until now. Recently, however, sunitinib and sorafenib showed its worth for NCRCC in extended access programs.1-3 Although it is not certain, the underlying mechanism of their action might lie in that papillary, chromophobe, and sarcomatoid type overexpress c-kit, which is also a target of both drugs and could therefore provide a therapeutic target for non-clear cell subtypes.4-7 Pazopanib is also a potent and selective, orally available, small molecule inhibitor of VEGFR-1,-2, and -3, PDGF-α, PDGF-β, and c-kit tyrosine kinases. It has been validated and licensed for advanced clear cell RCC (CCRCC).8 However, there is very few data about its efficacy for NCRCC.

In this study, we try to evaluate the efficacy of pazopanib in metastatic NCRCC.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 19 years
2. Subject must provide written informed consent
3. Histologically confirmed confirmation of renal cell carcinoma with more than 50% of a non clear cell histologic component:

   Include papillary type, chromophobe type, unclassified cell types; Exclude collecting duct and sarcomatoid type. (including sarcomatoid type or collecting duct type should be less than 5% in total cancer tumor)
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 -1
5. At least one measurable lesion by RECIST 1.1, which has not been affected previously with radiotherapy
6. Locally advanced or metastatic (stage IV) disease not amenable to surgery, radiotherapy, or combined modality therapy with curative intent
7. Subject who received immune therapy (interleukin-2, interferon) at least 6weeks time prior to the enrollment and at least 3 weeks time requires who received mTOR inhibitor (everolimus, temsirolimus) therapy prior to the enrollment.
8. Adequate organ system function as defined in the Table Definitions

   * Absolute neutrophil count (ANC):1.5 X 10^9/L
   * Hemoglobin: 9 g/dL (5.6 mmol/L)
   * Platelets: 100 X 10^9/L
   * Prothrombin time (PT) or international normalized ratio (INR):1.2 X ULN
   * Activated partial thromboplastin time (aPTT):1.2 X ULN
   * Total bilirubin:1.5 X ULN
   * Alanine amino transferase (ALT) and Aspartate aminotransferase (AST) should be in normal range in accordance with the site reference lab normal range
   * Serum creatinine: if >1.5 mg/dL: Calculated creatinine clearance (CIcr)≥30 mL/min
   * Urine Protein to Creatinine Ratio(UPC) <1 a. Blood transfusion is not allowed within 7days. b. Subject who takes anticoagulator therapy is eligible c. If urine protein to creatinine ratio is (UPC)≥1, must confirm the 24 hours urine and the protein should be <1g
9. A female is eligible to enter and participate in this study if she is of:

   1. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has had:

      • A hysterectomy
      * A bilateral oophorectomy (ovariectomy)
      * A bilateral tubal ligation
      * Is post-menopausal Subjects

        * not using hormone replacement therapy (HRT) must have experienced total cessation of menses for ≥ 1 year and be greater than 45 years in age, OR, in questionable cases, have a follicle stimulating hormone (FSH) value >40 mIU/mL and an estradiol value < 40pg/mL (<140 pmol/L).
        * Subjects using HRT must have experienced total cessation of menses for >= 1 year and be greater than 45 years of age OR have had documented evidence of menopause based on FSH and estradiol concentrations prior to initiation of HRT
   2. Childbearing potential, including any female who has had a negative serum pregnancy test within 2 weeks prior to the first dose of study treatment, preferably as close to the first dose as possible, and agrees to use adequate contraception. GSK acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follow:

      * Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product
      * Oral contraceptive
      * Injectable progestogen
      * Implants of levonorgestrel
      * Estrogenic vaginal ring
      * Percutaneous contraceptive patches
      * Intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1% per year
      * Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject
      * Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository) # Female subjects who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug.

Exclusion Criteria:

1. Patients who have 50% or more for component of clear cell type renal cell carcinoma
2. Prior malignancy cannot be included excepting for these cases: Subjects who have had another malignancy and have been disease-free for 2 years, or subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma and follicular or papillary thyroid cancer are eligible.
3. History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic for 4 weeks, and have had no requirement for steroids or anti-seizure medication for 2 weeks prior to first dose of study drug. Screening with CNS imaging studies (magnetic resonance imaging [MRI]) is required only if clinically indicated or if the subject has a history of CNS metastases.
4. Treatment with any of the following anti-cancer therapies:

   ① radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of pazopanib / RFA or cryoablation within 14 days prior to the first dose of pazopanib OR

   ② Prior treatment history with angiogenesis inhibitors such as sunitinib, sorafenib, bevacizumab is not permitted (prior MET inhibitor or c-kit inhibitor are also not permitted)

   ③ Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity, except alopecia.
5. Clinically significant gastrointestinal damage or disease that may affect absorption of pazopanib:

   (Active peptic ulcer disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or resection of the small bowel, history of stomy, abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28days prior to enrollment.)
6. Patients(male/female) of reproductive potential who are not use an effective contraceptive method
7. Pregnant, lactating women
8. Corrected QT interval (QTc) > 480 msecs
9. History of any severe disease or medical condition, significant heat failure(Class II, III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)) or pulmonary dysfunction, presence of uncontrolled active infection(requiring antibiotics)
10. History of clinically significant cardiac disease, arrhythmia and myocardial infarction
11. Symptomatic peripheral vascular disease
12. Poorly controlled hypertension [the patients who have systolic blood pressure (SBP) of <140 mmHg or diastolic blood pressure (DBP) of <90mmHg regardless antihypertensive treatment are eligible. If systolic blood pressure is 140-150mmHg, blood pressure (BP) must be re-assessed in a week and SBP <150mmHg is eligible.]
13. History of cerebrovascular accident including transient ischemic attack (TIA), untreated pulmonary embolism or deep venous thrombosis (DVT) within the past 2 months.
14. Prior major operation within 28 days prior to the first dose of study drug.
15. Evidence of active bleeding or bleeding diathesis.
16. Known lesions infiltrating major pulmonary vessels(simple abut lesion is eligible)
17. Hemoptysis in excess of 2.5 mL per cough (or one half teaspoon) due to cancer within 8 weeks of the first dose of study drug.
18. Unable or unwilling to discontinue use of prohibited medications listed in protocol for at least 14 days(whichever is longer) prior to the first dose of study drug and for the duration of the study.
19. Patients who are not capable of planned F/U visits due to pre-existing psychiatric, social and family condition or geographical reason.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-05-02 (Actual); Primary Completion 2015-02-28 (Actual); Study Completion 2015-11-14 (Actual)

PRIMARY OUTCOMES:
Overall response rates | 2years

SECONDARY OUTCOMES:
Progression-free survival | 2years
Overall survival | 2years
Number of Adverse Events | 2years
Exploratory analysis | 2years
  c-kit protein expression,the relationship between efficacy and tumoral fibroblast growth factor receptor 1 gene amplification (FISH), the relationship between efficacy and MET mutation in papillary carcinoma, the relationship between efficacy and microvessel density and/or VEGF-R2 expression in tumor by immunohistochemistry

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical Center, Seoul, South Korea